CLINICAL TRIAL: NCT02784886
Title: Cell-free Fetal DNA Circulating in the Maternal Plasma as a Marker for Morbidly Adherent Placenta in a High Risk Population
Brief Title: Cell-free Fetal DNA Circulating in the Maternal Plasma as a Marker for Morbidly Adherent Placenta
Acronym: DNA-Accreta
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: DC-2011-1467
Record Dates: First submitted 2016-05-19; First posted 2016-05-27 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Morbidly Adherent Placenta; Placenta Accreta; Placenta Increta; Placenta Percreta
Keywords: Placenta accreta; previous caesarean; placenta praevia; Cell-free fetal DNA; Biological markers
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Women at high risk of MAP — Blood sample

SUMMARY:
The purpose of this study is to determine whether, in a high risk population (placenta praevia and previous caesarean or prenatal suspicion of morbidly adherent placenta (MAP)), the concentration of cell-free fetal DNA circulating in the maternal plasma is significantly increased in the subgroup of morbidly adherent placenta (MAP) cases , in order to determine if the dosage of cell-free fetal DNA circulating in the maternal plasma may be a useful biological tool to detect MAP, alone or in addition to the imagery findings (ultrasonography and RMI).

DETAILED DESCRIPTION:
Background: Morbidly adherent placenta (MAP) is a life-threatening condition characterized by placental villi being abnormally adherent to the myometrium. Prenatal identification of MAP is essential to anticipate the risk and plan optimal delivery conditions for these women while this is associated to a maternal outcome improvement. Prenatal identification based on Doppler ultrasound and/or MRI is associated with high rates of false-positive or false-negative findings responsible for adverse effects. Some cases reports have suggested that the concentration of cell-free fetal DNA circulating in the maternal plasma is significantly increased in a context of morbidly adherent placenta (MAP).

Objective: The primary objective is to determine whether the concentration of cell-free fetal DNA circulating in the maternal plasma is significantly increased in women with morbidly adherent placenta (MAP) compared to women with placenta praevia and previous caesarean. Secondary objectives are to determine whether cell-free fetal DNA circulating in the maternal plasma is a useful biological tool to detect MAP, alone or in addition to the imagery findings (ultrasonography and RMI), in a high risk population (placenta praevia and previous caesarean or only prenatal suspicion of MAP).

Design: Prospective observational study of pregnant women with placenta praevia and previous cesaeran or with prenatal suspicion of placenta accreta, conducted in 5 centers.

Methods: We expect to include 83 women at risk of MAP in two years, of whom approximately 17 (20%) will have a MAP.

Main outcome measures: The primary outcome measure is concentration of cell-free fetal DNA circulating in maternal plasma.

Conclusion: This study will be the first prospective study to include women at risk of placenta accreta and to investigate whether the concentration of cell-free fetal DNA circulating in maternal plasma is increased in MAP women and whether it is a useful biological marker to detect prenatally MAP in a high risk population.

ELIGIBILITY:
Inclusion Criteria:

Every woman:

* delivering in one of the 5 maternity units that participate to a Population-based prospective observational study of pregnant women with a placenta praevia and previous cesarean or with prenatal suspicion of accreta (PACCRETA) .
* With a placenta praevia and at least one previous cesarean delivery or having a prenatal suspicion of placenta accreta
* aged 18 or more

Exclusion Criteria:

Every woman:

* not understanding French.
* refusing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women delivering in 5 maternity units that participate in a Population-based prospective observational study of pregnant women with a placenta praevia and previous cesarean or with prenatal suspicion of accreta (PACCRETA)
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2013-11; Primary Completion 2015-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Concentration of cell-free fetal DNA circulating in the maternal plasma | from 24 weeks gestation to delivery

SECONDARY OUTCOMES:
Sensitivity of the concentration of cell-free fetal DNA | from 24 weeks gestation to delivery
Specificity of the concentration of cell-free fetal DNA | from 24 weeks gestation to delivery
Positive predictive value of concentration of cell-free fetal DNA | from 24 weeks gestation to delivery
Negative predictive value of the concentration of cell-free fetal DNA | from 24 weeks gestation to delivery
Sensitivity, specificity, positive predictive value (PPV) and negative (NPV) of the concentration of cell-free fetal DNA in association with clinical criteria ( risk factors for MAP) | from 24 weeks gestation to delivery
Sensitivity, specificity, positive predictive value (PPV) and negative (NPV) of concentration of cell-free fetal DNA in association with imaging criteria magnetic resonance | from 24 weeks gestation to delivery
Sensitivity, specificity, positive predictive value (PPV) and negative (NPV) of the concentration of cell-free fetal DNA and clinical criteria in association with clinical criteria, sonographic criteria and with magnetic resonance imaging criteria | from 24 weeks gestation to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Deneux-Tharaux, MD, PhD, Study Director — Inserm U1153, Obstetrical, Perinatal and Pediatric Epidemiology Research Team, Paris, France
Locations (1):
- Angers University Hospita, Angers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sekizawa A, Jimbo M, Saito H, Iwasaki M, Sugito Y, Yukimoto Y, Otsuka J, Okai T. Increased cell-free fetal DNA in plasma of two women with invasive placenta. Clin Chem. 2002 Feb;48(2):353-4. No abstract available. PMID 11805017
- [Background] Jimbo M, Sekizawa A, Sugito Y, Matsuoka R, Ichizuka K, Saito H, Okai T. Placenta increta: Postpartum monitoring of plasma cell-free fetal DNA. Clin Chem. 2003 Sep;49(9):1540-1. doi: 10.1373/49.9.1540. No abstract available. PMID 12928242
- [Background] Kayem G, Deneux-Tharaux C, Sentilhes L; PACCRETA group. PACCRETA: clinical situations at high risk of placenta ACCRETA/percreta: impact of diagnostic methods and management on maternal morbidity. Acta Obstet Gynecol Scand. 2013 Apr;92(4):476-82. doi: 10.1111/aogs.12078. Epub 2013 Feb 15. PMID 23360123
- [Background] Sentilhes L, Goffinet F, Kayem G. Management of placenta accreta. Acta Obstet Gynecol Scand. 2013 Oct;92(10):1125-34. doi: 10.1111/aogs.12222. PMID 23869630